CLINICAL TRIAL: NCT06389617
Title: Different Doses of Intravenous Administered Dexamethasone Effecting Brachial Plexus Supraclavicular Block for Creation of Arteriovenous Fistula in End Stage Renal Disease: A Randomized Controlled Trial
Brief Title: Different Doses of Intravenous Administered Dexamethasone Effecting Brachial Plexus Supraclavicular Block
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Prem Anand A/L Tb Nantha Kumar, Dr, Hospital Universiti Sains Malaysia
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: USM/JEPeM/KK/24010061
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: End Stage Renal Failure
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GROUP DF (Active Comparator): supraclavicular block with 20mls of Ropivacaine 0.5% and Intravenous dexamethasone 4mg
  Interventions: Drug: supraclavicular block with 20mls of Ropivacaine 0.5% and Intravenous administered dexamethasone
- GROUP DE (Active Comparator): supraclavicular block with 20mls of Ropivacaine 0.5% and Intravenous dexamethasone 8mg
  Interventions: Drug: supraclavicular block with 20mls of Ropivacaine 0.5% and Intravenous administered dexamethasone

INTERVENTIONS:
Drug: supraclavicular block with 20mls of Ropivacaine 0.5% and Intravenous administered dexamethasone — Comparing the onset of sensory, motor block, duration of motor block and analgesic duration

SUMMARY:
To compare the analgesic properties of ultrasound guided supraclavicular block using ropivacaine 0.5% in arteriovenous fistula creation when used in combination with intravenous administered dexamethasone at 4mg and 8 mg as an adjuvant

ELIGIBILITY:
Inclusion Criteria:

Adult, age 18 to 65 years End stage renal disease patients for AV fistula creation

Exclusion Criteria:

Not suitable candidate as determined by the primary team Refusal for brachial plexus block History of allergy to dexamethasone or local anesthesia Pregnancy History of previous brachial plexus injury Coagulopathy Local skin site infection Known neuropathy involving the arm undergoing surgery Patients with glucose reading more then 12mmol/

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
To compare the difference of onset time between sensory and motor block of supraclavicular block between ropivacaine with IV dexamethasone 4mg and ropivacaine with IV dexamethasone 8mg | 2 days
To compare the difference in duration of analgesia between supraclavicular block with ropivacaine and IV dexamethasone 4mg with ropivacaine and IV dexamethasone 8mg | 2 days

SECONDARY OUTCOMES:
To compare the duration difference of the return of motor block between supraclavicular block using ropivacaine with IV dexamethasone 4mg and ropivacaine with IV dexamethasone 8mg | 2 days